CLINICAL TRIAL: NCT07093164
Title: Randomized Controlled Single-blind Non-inferiority Trial Comparing an Offer of Initial Virtual Visit and Usual Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Deemed infeasible.
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, Professor of surgery and perioperative care, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-11-0170
Record Dates: First submitted 2020-02-01; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Musculoskeletal Diseases
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: . Patients will be randomized using a random number generator in Microsoft Excel in 1:1 ratio to a standard in person visit OR to be called by a research assistant to offer a virtual visit in advance of an in person visit. Patients that indicate interest in a virtual visit will make a scheduled video appointment and test the website to be used in conjunction with the research assistant.
  At the end of the virtual visit, if patients decide to cancel the in person visit, they will be asked to complete a REDCap survey via text link.
Who Masked: Participant
Masking Description: We will request a waiver of informed consent in order to blind the patients for this trial. As initial visits already take place both in person and virtual, we do not feel the blinding or randomization adds risk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In person visit (No Intervention): Patients will be provided an initial in person visit. Patients that visit in person will complete the REDCap survey after the visit.
- Virtual visit (Experimental): Patients will be provided an initial virtual health or telehealth visit. At the end of the virtual visit, if patients decide to cancel the in person visit, they will be asked to complete a REDCap survey via text link.
  Interventions: Behavioral: Virtual visit

INTERVENTIONS:
Behavioral: Virtual visit — Patients will be provided an initial virtual health or telehealth visit instead of an in person visit.
  Arms: Virtual visit

SUMMARY:
This randomized controlled trial will address whether there is a difference in satisfaction with treatment plan, satisfaction with the clinician, perceived empathy, patient reported outcomes, and psychological measures among patients randomized to the offer of an initial virtual health or telehealth visit compared to those provided an initial in person visit.

DETAILED DESCRIPTION:
Virtual visits (video) provide people seeking care additional options. The quality of virtual care resources has improved, making it a user-friendly way to address health concerns. The benefits of virtual visits include no travel time, less time away from work, and no need for dependent care arrangements.

Previous studies found virtual visits to be safe, efficient and accurate for selected orthopaedic patients . An RCT found telemedicine capable of providing a satisfactory standard care in the management of minor injuries. Others suggest that virtual care is an alternative to in person visits for orthopaedic patients in an outpatient setting.

There are concerns that virtual care will represent another commodity that will increase the amount and costs of care without increasing health as was observed for retail care. On the other hand, there is evidence that online care for simple conditions saves money. Also a pilot study showed that online visits appeared to reduce medical costs for patients during a 6-month period after the visit.

This randomized controlled trial will address whether there is a difference in satisfaction with treatment plan, satisfaction with the clinician, perceived empathy, patient reported outcomes, and psychological measures among patients randomized to the offer of an initial virtual health or telehealth visit compared to those provided an initial in person visit.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Between 17 and 90 years old
* musculoskeletal problem
* New and returned

Exclusion Criteria:

-

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Guttman Satisfaction scale | At time of initial visit and again 1 month following visit
  The Guttman Satisfaction Scale is a unidimensional questionnaire designed to measure the degree of patient satisfaction with the care they received. It consists of a series of hierarchically ordered yes/no items, with each successive item indicating a higher level of satisfaction. Total scores range from 0 to 7, with higher scores reflecting greater satisfaction, representing a better outcome.

SECONDARY OUTCOMES:
Jefferson scale of patient perception of physician empathy | Once only - after initial visit
  The Jefferson Scale of Patient's Perceptions of Physician Empathy includes five items rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree), with total scores ranging from 5 to 35. Higher scores indicate greater perceived physician empathy, representing a better outcome.
Patient Reported Outcome Measurement Information System(PROMIS) Upper extremity Physical Function Computer Adaptive Test | At time of initial visit and again 1 month following visit
  Patient physical function will be assessed using the PROMIS Upper Extremity Computer Adaptive Test (CAT). This instrument evaluates the ability to perform daily activities requiring upper limb function, such as reaching, lifting, and fine motor tasks. Scores are reported as T-scores, ranging from 20 (indicating minimum physical ability) to 80 (maximum physical ability). Higher scores reflect better upper extremity function and therefore a better outcome.
Pain intensity scale | At time of initial visit and again 1 month following visit
  Pain intensity will be assessed using a numerical rating scale ranging from 0 to 10, where 0 indicates "no pain" and 10 indicates "the worst pain imaginable." Higher scores reflect greater pain intensity and therefore a worse outcome.
Number of diagnostic tests or treatments | Cumulative total at 1 month following visit)
  Total number of all tests or treatments performed for patient, including: injections, imaging studies and procedures.

OTHER OUTCOMES:
Short Health Anxiety Inventory 5 (SHAI-5) | Once only (at time of initial visit)
  The Short Health Anxiety Inventory 5-item version (SHAI-5) is a brief questionnaire designed to assess health-related anxiety. Each item is rated on a 4-point scale (0 to 3), with total scores ranging from 0 to 15. Higher scores indicate greater health anxiety.
Pain Catastrophizing Scale (PCS-4) | Once only (at time of initial visit)
  The Pain Catastrophizing Scale - 4 item version (PCS-4) is a mental health measure assessing the extent of catastrophic thoughts related to pain. It consists of 4 items rated on a 5-point scale (0 = not at all to 4 = all the time), with total scores ranging from 0 (no pain catastrophizing) to 16 (highest level of pain catastrophizing). Higher scores indicate greater catastrophic thinking.
Patient Health Questionnaire (PHQ-2) | Once only (at time of initial visit)
  The Patient Health Questionnaire-2 (PHQ-2) is a brief mental health screening tool measuring the frequency of core depressive symptoms over the past two weeks. It includes 2 items scored from 0 ("not at all") to 3 ("nearly every day"), with total scores ranging from 0 (no depressive symptoms) to 6 (highest level of depressive symptoms). Higher scores indicate greater severity of depressive symptoms, representing a worse outcome.

IPD SHARING:
Plan to Share IPD: No